CLINICAL TRIAL: NCT01890291
Title: Long Term Study of 'Immuncell-LC Groups' and 'Non-treatment Groups' in Patient Undergo Curative Resection (PEIT, Radiofrequency Ablation [RFA] or Operation) for Hepatocellular Carcinoma in Korea
Brief Title: Long Term Follow-Up Study of Immuncell-LC Group and Non-Treatment Group in Hepatocellular Carcinoma Patients.
Acronym: Immuncell-LC
Status: Completed | Type: Observational
Sponsor: GC Cell Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: IIC-I02
Record Dates: First submitted 2013-06-24; First posted 2013-07-01 (Estimated); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Immuncell-LC, Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-treatment Group: Patients who were in non-treatment group in phase 3 clinical trial IIC-I01(NCT00699816).
- Immuncell-LC Group: Patients who were in Immuncell-LC group in phase 3 clinical trial IIC-I01(NCT00699816).

SUMMARY:
To observation that long term follow-up study of 'Immuncell-LC groups' and 'Non-treatment groups' in patient undergo curative resection (PEIT, RFA or Operation) for hepatocellular carcinoma in Korea

ELIGIBILITY:
Inclusion Criteria:

* Prior to the test, patient is fully explained about the purpose/ contents and characteristics of the testing medication, and the patient him(her)self, the guardian or the legal representative signed on written consent.
* Patients of participated in the(ClinicalTrials.gov Identifier:NCT00699816)clinical trial.

Exclusion Criteria:

* Patient who is incongruent to this clinical trial by sub-investigator's opinion.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This long term follow-UP study is observation about the Immuncell-LC Groups' and 'Non-treatment Groups' in patient undergo curative resection (PEIT, RFA or Operation) for Hepatocelluar Carcinoma in Korea.
Sampling Method: Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2013-06; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
To evaluate recurrence-free survival | up to 3 years
  Radiological test should be operated by dynamic CT(using 64 cut), dynamic MRI or by angiography.

SECONDARY OUTCOMES:
To determine the response rate to evaluate overall survival and cause specific survival and changes of Alpha feto protein (AFP) figures from baseline to the last observation date. | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jung Hwan Yoon, MD, Principal Investigator — Seoul National University Hospital; Joon Hyeok Lee, MD, Principal Investigator — Samsung Medical Center; Young-Suk Lim, MD, Principal Investigator — Asan Medical Center; Tae Gin Song, MD, Principal Investigator — Korea University Ansan Hospital; Jong Eun Yeon, MD, Principal Investigator — Korea University Guro Hospital
Locations (5):
- South Korea (5):
  - Seoul National Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Korea University Ansan Hospital, Seoul